CLINICAL TRIAL: NCT05071716
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Rifaximin Soluble Solid Dispersion (SSD) for the Delay of Encephalopathy Decompensation in Cirrhosis
Brief Title: Study to Assess Rifaximin Soluble Solid Dispersion (SSD) for the Delay of Encephalopathy Decompensation in Cirrhosis
Acronym: RED-C-3131
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RNLC3131
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifaximin SSD-40mg IR (Experimental)
  Interventions: Drug: Rifaximin SSD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin SSD — Rifaximin Solid Soluble Dispersion Immediate Release Twice Daily
  Arms: Rifaximin SSD-40mg IR
Drug: Placebo — Placebo Twice Daily
  Arms: Placebo

SUMMARY:
Study RNLC3131 is a Phase 3, randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of rifaximin SSD-40mg IR for the delay of the first episode of overt hepatic encephalopathy (OHE) decompensation in liver cirrhosis, defined by the presence of medically controlled ascites.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of liver cirrhosis with medically controlled ascites (>30 days) not requiring therapeutic paracentesis (could have had paracentesis in the past).
* Conn (West Haven Criteria) score of < 2.
* Mini-Mental State Examination (MMSE) score > 24 at screening.
* ≥ 18 and ≤ 85 years of age.

Key Exclusion Criteria:

* Active COVID-19 that is unresolved
* History of SBP
* History of EVB or AKI-HRS within 6 months
* History of OHE episode (Conn score ≥ 2)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Time to first event of overt hepatic encephalopathy requiring medical intervention in hospital/ER/ED/clinic or death. | 72 weeks

SECONDARY OUTCOMES:
Time to first Conn score ≥ 2 or confirmed OHE requiring medical intervention in hospital/ER/ED/ clinic or death | 72 weeks
Time to all-cause hospitalization | 72 weeks
Time to first event of OHE that requires hospitalization, or all-cause death | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mader, Study Director — Bausch Health
Locations (150):
- United States (139):
  - Bausch Site 182, Dothan, Alabama
  - Bausch Site 129, Chandler, Arizona
  - Bausch Site 103, Peoria, Arizona
  - Bausch Site 180, Phoenix, Arizona
  - Bausch Site 153, Phoenix, Arizona
  - Bausch Site 248, Tempe, Arizona
  - Bausch Site 222, Tucson, Arizona
  - Bausch Site 150, Little Rock, Arkansas
  - Bausch Site 164, Bakersfield, California
  - Bausch Site 196, Chula Vista, California
  - Bausch Site 226, Chula Vista, California
  - Bausch Site 174, Escondido, California
  - Bausch Site 163, Fresno, California
  - Bausch Site 242, Garden Grove, California
  - Bausch Site 115, La Jolla, California
  - Bausch Site 141, Lancaster, California
  - Bausch Site 140, Los Angeles, California
  - Bausch Site 189, Los Angeles, California
  - Bausch Site 227, Orange, California
  - Bausch Site 199, Pasadena, California
  - Bausch Site 119, Redwood City, California
  - Bausch Site 102, Rialto, California
  - Bausch Site 177, San Diego, California
  - Bausch Site 171, San Francisco, California
  - Bausch Site 214, San Jose, California
  - Bausch Site 183, Upland, California
  - Bausch Site 143, Englewood, Colorado
  - Bausch Site 212, Littleton, Colorado
  - Bausch Site 151, Bristol, Connecticut
  - Bausch Site 220, Bradenton, Florida
  - Bausch Site 257, Cape Coral, Florida
  - Bausch Site 197, Cutler Bay, Florida
  - Bausch Site 249, Fort Myers, Florida
  - Bausch Site 173, Hialeah, Florida
  - Bausch Site 238, Hialeah Gardens, Florida
  - Bausch Site 235, Hollywood, Florida
  - Bausch Site 211, Homestead, Florida
  - Bausch Site 139, Inverness, Florida
  - Bausch Site 138, Jacksonville, Florida
  - Bausch Site 241, Lakewood Rch, Florida
  - Bausch Site 157, Miami, Florida
  - Bausch Site 255, Miami, Florida
  - Bausch Site 263, Miami, Florida
  - Bausch Site 264, Miami, Florida
  - Bausch Site 268, Miami, Florida
  - Bausch Site 224, Miami, Florida
  - Bausch Site 243, Miami, Florida
  - Bausch Site 166, Miami, Florida
  - Bausch Site 244, Miami, Florida
  - Bausch Site 266, Miami, Florida
  - Bausch Site 147, Miami, Florida
  - Bausch Site 218, Miami, Florida
  - Bausch Site 240, Miami, Florida
  - Bausch Site 186, New Port Richey, Florida
  - Bausch Site 213, Orlando, Florida
  - Bausch Site 267, Pembroke Pines, Florida
  - Bausch Site 256, Plantation, Florida
  - Bausch Site 272, Venice, Florida
  - Bausch Site 188, Weston, Florida
  - Bausch Site 219, Atlanta, Georgia
  - Bausch Site 215, Augusta, Georgia
  - Bausch Site 260, Dalton, Georgia
  - Bausch Site 126, Marietta, Georgia
  - Bausch Site 194, Chicago, Illinois
  - Bausch Site 120, Indianapolis, Indiana
  - Bausch Site 152, Clive, Iowa
  - Bausch Site 135, Iowa City, Iowa
  - Bausch Site 128, Topeka, Kansas
  - Bausch Site 124, Louisville, Kentucky
  - Bausch Site 237, Baton Rouge, Louisiana
  - Bausch Site 261, Houma, Louisiana
  - Bausch Site 134, Marrero, Louisiana
  - Bausch Site 118, New Orleans, Louisiana
  - Bausch Site 117, Baltimore, Maryland
  - Bausch Site 230, Glen Burnie, Maryland
  - Bausch Site 132, Boston, Massachusetts
  - Bausch Site 161, Boston, Massachusetts
  - Bausch Site 223, Boston, Massachusetts
  - Bausch Site 146, Burlington, Massachusetts
  - Bausch Site 233, New Bedford, Massachusetts
  - Bausch Site 136, Ann Arbor, Michigan
  - Bausch Site 265, Detroit, Michigan
  - Bausch Site 137, Detroit, Michigan
  - Bausch Site 149, Wyoming, Michigan
  - Bausch Site 253, Minneapolis, Minnesota
  - Bausch Site 271, Minneapolis, Minnesota
  - Bausch Site 148, Jackson, Mississippi
  - Bausch Site 178, Kansas City, Missouri
  - Bausch Site 251, East Brunswick, New Jersey
  - Bausch Site 191, Newark, New Jersey
  - Bausch Site 216, Albuquerque, New Mexico
  - Bausch Site 109, New York, New York
  - Bausch Site 225, New York, New York
  - Bausch Site 116, New York, New York
  - Bausch Site 217, Charlotte, North Carolina
  - Bausch Site 192, Durham, North Carolina
  - Bausch Site 269, Statesville, North Carolina
  - Bausch Site 245, Wilmington, North Carolina
  - Bausch Site 273, Wilmington, North Carolina
  - Bausch Site 114, Cleveland, Ohio
  - Bausch Site 154, Columbus, Ohio
  - Bausch Site 167, Dayton, Ohio
  - Bausch Site 185, Mentor, Ohio
  - Bausch Site 270, Moore, Oklahoma
  - Bausch Site 110, Philadelphia, Pennsylvania
  - Bausch Site 228, Pittsburgh, Pennsylvania
  - Bausch Site 250, Sayre, Pennsylvania
  - Bausch Site 104, Charleston, South Carolina
  - Bausch Site 184, Johnson City, Tennessee
  - Bausch Site 181, Nashville, Tennessee
  - Bausch Site 221, Austin, Texas
  - Bausch Site 122, Dallas, Texas
  - Bausch Site 144, Dallas, Texas
  - Bausch Site 133, Dallas, Texas
  - Bausch Site 107, Dallas, Texas
  - Bausch Site 123, Denison, Texas
  - Bausch Site 198, El Paso, Texas
  - Bausch Site 172, Fort Worth, Texas
  - Bausch Site 210, Fort Worth, Texas
  - Bausch Site 258, Harlingen, Texas
  - Bausch Site 170, Houston, Texas
  - Bausch Site 130, Houston, Texas
  - Bausch Site 158, Houston, Texas
  - Bausch Site 159, Houston, Texas
  - Bausch Site 229, Houston, Texas
  - Bausch Site 239, Houston, Texas
  - Bausch Site 252, Mesquite, Texas
  - Bausch Site 195, Pearland, Texas
  - Bausch Site 247, Sugar Land, Texas
  - Bausch Site 262, Sugar Land, Texas
  - Bausch Site 246, Texas City, Texas
  - Bausch Site 193, Waco, Texas
  - Bausch Site 127, Murray, Utah
  - Bausch Site 231, Manassas, Virginia
  - Bausch Site 175, Norfolk, Virginia
  - Bausch Site 113, Richmond, Virginia
  - Bausch Site 111, Richmond, Virginia
  - Bausch Site 155, Seattle, Washington
  - Bausch Site 105, Milwaukee, Wisconsin
- Australia (7):
  - Bausch Site 307, Concord, New South Wales
  - Bausch Site 300, Kingswood, New South Wales
  - Bausch Site 306, Bedford Park, South Australia
  - Bausch Site 304, Box Hill, Victoria
  - Bausch Site 302, Parkville, Victoria
  - Bausch Site 305, Murdoch, Western Australia
  - Bausch Site 303, Perth, Western Australia
- Canada (3):
  - Bausch Site 202, Edmonton, Alberta
  - Bausch Site 203, Toronto, Ontario
  - Bausch Site 201, Toronto, Ontario
- Bausch Site 234, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180